CLINICAL TRIAL: NCT05897034
Title: Clinical Study to Investigate the Effect of Doxycycline, Pentoxifylline, and Nitazoxanide in Sexually Active Men
Brief Title: Combination Therapy Between Doxycycline, Pentoxifylline, and Nitazoxanide in Sexually Active Men
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Mostafa Mahmoud Bahaa Clinical Pharmacy Department, Horus University, New Damietta, Egypt (Unknown)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching assisstant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3568
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Doxycycline; Pentoxifylline; nitazoxanide; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): This group will take doxycycline 100 mg twice daily
  Interventions: Drug: Doxycyclin
- Comparative group (Active Comparator): This group will take doxycycline 100 mg twice daily, pentoxifylline 400 mg twice daily, and nitazoxanide 500 mg twice daily.
  Interventions: Drug: Doxycyclin; Drug: Pentoxifylline; Drug: Nitazoxanide 500Mg Oral Tablet

INTERVENTIONS:
Drug: Doxycyclin — Doxycycline is a moderate-spectrum, second-generation tetracycline that is generally well tolerated
Drug: Pentoxifylline — Pentoxifylline is a vasoactive agent that improves the flow of blood by reducing its viscosity
  Arms: Comparative group
Drug: Nitazoxanide 500Mg Oral Tablet — Nitazoxanide is a broad-spectrum antiparasitic and broad-spectrum antiviral medication that is used in medicine for the treatment of various helminthic, protozoal, and viral infections
  Arms: Comparative group

SUMMARY:
Bacterial sexually transmitted infections (STIs) have been steadily increasing in gay, bisexual, and other men who have sex with men (MSM) over the past 2 decades. While that trend started prior to the introduction of human immunodeficiency virus (HIV) pre-exposure prophylaxis (PrEP) in 2012, HIV PrEP has been associated with increases in sexual contacts and decreases in condom use with an resultant acceleration in the increase of bacterial STIs such as gonorrhea, syphilis, and chlamydia.

DETAILED DESCRIPTION:
Doxycycline is a moderate-spectrum, second-generation tetracycline that is generally well tolerated. It is rapidly and almost completely absorbed after oral administration. First introduced commercially in the 1960s, doxycycline has been used by millions to manage acne and as primary prophylaxis for scrub typhus, leptospirosis, malaria, and Lyme disease. There are anecdotal reports of doxycycline used for syphilis prophylaxis among US and Australian military personnel during the Vietnam War. Doxycycline is a first-line agent for treatment of chlamydia and an alternative regimen for syphilis.An open-label extension of the French national HIV research agency (France Recherche Nord & sud Sida-hiv hépatites [ANRS]) Intervention Préventive de l'Exposition aux Risques avec et pour les Gays (IPERGAY) HIV-prevention study continued participant access to HIV PrEP and examined doxycycline postexposure prophylaxis (Doxy PEP) in MSM and transgender women without HIV [17]. Participants (n = 232) were randomly assigned 1:1 to the intervention-doxycycline 200 mg within 24-72 hours of condomless sexual encounters up to 3 times per week-or to no prophylaxis. Those taking Doxy PEP had lower STI incidence (hazard ratio, 0.57; P = .014). Chlamydia trachomatis and syphilis diagnoses were significantly lower in the intervention arm, with a relative reduction of 70-73% in the intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged > 18 years were eligible for participation if they had a diagnosis of untreated gonorrhea and chlamydia. The untreated status was defined as no antibiotic taken in the previous 28 days to treat gonorrhea and chlamydia.

Exclusion Criteria:

* known contraindications or hypersensitivity to doxycycline, pentoxifylline, and nitazoxanide.

gonorrhea with complications, such as pelvic inflammatory disease or epididymo-orchitis significant renal failure or hepatic failure.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2024-06-20 (Estimated); Study Completion 2028-06-20 (Estimated)

PRIMARY OUTCOMES:
treatment of chylamdia in sexually active men | 1 month
  treatment of chylamdia in sexually active men and decreasing resistance to antibiotics